CLINICAL TRIAL: NCT03828903
Title: The Diagnostic Value of Cryobiopsy During Medical Thoracoscopy in Diagnosis of Pleural Effusion
Brief Title: Role of Cryobiopsy in Diagnosis of Pleural Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Salah Abd El Ghany, Assistant lecturer, Chest Department and tuberculosis, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cryobiopsy pleural effusion
Record Dates: First submitted 2019-01-26; First posted 2019-02-04 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-10

CONDITIONS: Pleural Effusion
Keywords: Cryobiopsy
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pleural effusion patients (Experimental): medical thoracoscopy will e performed to patients with pleural effusion and pleural biopsy by forceps ad cryoprobe will be obtained
  Interventions: Device: Cryoprobe

INTERVENTIONS:
Device: Cryoprobe — * The probe (ERBE Elektromedizin GmbH; Tubingen, Germany of 2.4mm) will be placed perpendicular to the surface of the parietal pleura with the tip of the probe extended well beyond the tip of the scope using the marking on the probe and with direct visualization.
  * The tip of the cryoprobe will be attached to suspicious part of parietal pleura .
  * The frozen tissue is going to be extracted by gently pulling of the probe.
  * Freezing will be carried out for 6 to 10 seconds depending on the visual assessment of pleural texture.
  * The probe with the attached biopsy sample is going to be removed together with the thoracoscope through trocar.
  * The biopsy sample will be released from the probe by thawing in the saline.
  * The semirigid pleuroscope will be reintroduced through the port and the pleura will be revisualized for bleeding.

SUMMARY:
The purpose of this study is to evaluate the feasibility, size and quality of the specimens obtained by cryoprobe in comparison to those specimens obtained by flexible forceps during medical thoracoscopy in diagnosis of pleural effusion.

DETAILED DESCRIPTION:
* Medical thoracoscopy with single-port-of-entry technique will be performed in the bronchoscopy unit under local anesthesia and conscious sedation using midazolam (2 mg) or pethidin.
* vertical incision will be made with the scalpel (usually near the midaxillary line), through the skin and subcutaneous tissue, appropriate to the size of the trocar to be used, usually of approximately 10 mm, parallel with and in the middle of the selected intercostal space.
* Then the trocar will be inserted until the sudden release of resistance (after passing the costal pleura) is felt.
* Under direct vision with the thoracoscope, introduction of pneumothorax will be performed, and all pleural fluid will be removed, and the pleural cavity will be inspected.
* Suspicious areas will be biopsied through the working channel of the thoracoscope.
* two to six biopsies of a suspicious pleural lesion will establish the diagnosis.

Technique of pleural biopsy using cryotechnique:

* The probe (ERBE Elektromedizin GmbH( Gesellschaft mit beschränkter Haftung) , Germany of 2.4mm) will be placed perpendicular to the surface of the parietal pleura with the tip of the probe extended well beyond the tip of the scope using the marking on the probe and with direct visualization.
* The tip of the cryoprobe will be attached to suspicious part of parietal pleura and activated by footswitch.
* carbon dioxide will be used as the cryogen gas for cryobiopsy
* The frozen tissue is going to be extracted by gently pulling of the probe.
* Freezing will be carried out for 6 to 10 seconds depending on the visual assessment of pleural texture.

ELIGIBILITY:
Inclusion Criteria:

- 1. Unilateral moderate or massive exudative pleural effusion patients. 2. Undiagnosed pleural effusion after simple pleural fluid aspiration, cytology or blind (closed) pleural biopsy using Abram's needle.

3. Age>18 years old

Exclusion Criteria:

1. Transudative pleural effusion.
2. Exudative pleural effusion less than one third of hemithorax.
3. Presence of hemorrhagic diathesis (prothrombin concentration <50% and platelet count <80,000/mm 3).
4. Poor performance state (ECOG performance status >4) as recommended in BTS (British thoracic society) guidelines 2010.
5. Sever uncontrollable cough, hypercapnia and sever respiratory distress.
6. Fibrothorax, excessive pleural adhesion.

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
comparison between pleural biopsy specimens obtained by flexible forceps with those obtained with cryoprobe during medical thoracoscopy in diagnosis of pleural effusion. | 12 months
  1_size of pleural biopsy obtained by cryoprobe in comparison to those obtained by flexible forceps (in millimeter).

SECONDARY OUTCOMES:
Complication assessment | 12 months
  To evaluate the safety and occurrence of complication such as bleeding Number of patients with a certain degree of bleeding from biopsy site, described as:
  1 = slight, self-limited, 2 = moderate, requiring electrocautery intervention, 3 = severe, requiring interruption of the procedure, chest tube drainage and intravenous fluid resuscitation .
assessment pleural fluid | 12 months
  comparison between the estimate of pleural effusion using chest ultrasound and actual amount after thoracoscpic drainage, measured in mililiters.
assessment of post procedure pain | 12 months
  comparison between meperidine and (midazolam &NSAIDs) in controlling pain post thoracoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Reham M El morshedy, Lecturer, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Assuit University hospital, Asyut
  - Alaa Salah Abdel gany, Asyut

REFERENCES:
- [Background] Chen CH, Cheng WC, Wu BR, Chen CY, Chen WC, Liao WC, Tu CY. Feasibility and Safety of Pleuroscopic Cryobiopsy of the Pleura: A Prospective Study. Can Respir J. 2018 Jan 22;2018:6746470. doi: 10.1155/2018/6746470. eCollection 2018. PMID 29610630
- [Background] Tousheed SZ, Manjunath PH, Chandrasekar S, Murali Mohan BV, Kumar H, Hibare KR, Ramanjaneya R. Cryobiopsy of the Pleura: An Improved Diagnostic Tool. J Bronchology Interv Pulmonol. 2018 Jan;25(1):37-41. doi: 10.1097/LBR.0000000000000444. PMID 29261578